CLINICAL TRIAL: NCT05240313
Title: Preventing Alcohol and Other Drug Use and Violence Among Latino Youth
Acronym: kiR-vene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christopher Salas-Wright, Professor, Boston College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5110411; 5K01AA026645-05 (NIH)
Record Dates: First submitted 2022-01-21; First posted 2022-02-15 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Drinking; Violence in Adolescence
Keywords: Latino; Adolescent; Immigrant
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- keepin' it REAL (kiR) (Experimental): The standard keepin' it REAL intervention, adapted for an online format. This includes 10 one-hour small group sessions focused on helping youth to develop drug refusal skills and improve decision making, risk assessment, and emotion regulation. Additionally, short videos highlight various aspects of the program (refuse, explain, avoid, leave). All materials are available in Spanish and English.
  Interventions: Behavioral: kiR venezolano
- kiR + aggression (Experimental): The standard keepin' it REAL intervention, adapted for an online format, plus content on interpersonal aggression
  Interventions: Behavioral: kiR venezolano
- Stress Management (Active Comparator): A single session focused on stress management skills.
  Interventions: Behavioral: kiR venezolano

INTERVENTIONS:
Behavioral: kiR venezolano — A multi-week intervention focused on drug refusal skills and self-regulation.

SUMMARY:
There are currently no interventions aimed at preventing both alcohol and other drug (AOD) use and interpersonal violence that have been adapted for Latino adolescents. This study hypothesizes that a cultural adaptation of a validated AOD use prevention program (Keepin' it REAL) that also integrates violence prevention content will both amplify the AOD use effects of that intervention for Latino adolescents and lead to reductions in youth violence.

The purpose of this study is to conduct a pilot-test randomized controlled trial (RCT) of a youth AOD use prevention intervention that has been adapted to integrate interpersonal violence content and has been culturally adapted for a specific Latino population (Venezuelan migrant youth). The goals of the pilot test are to determine feasibility, acceptability, and preliminary effects of the intervention for future testing.

DETAILED DESCRIPTION:
The intervention will be an adaptation of Keepin' it REAL (KiR). KiR is a 10-week intervention for early adolescents that is considered a model evidence-based AOD use prevention program by SAMHSA. It based on communications theory and the importance of aligning cultural values with AOD outcomes. Weekly sessions focus on teaching youth communications strategies to enhance their ability to navigate situations where substance use may be present. It incorporates a student workbook, videos, and in-session discussions and exercises. We will be adapting the intervention for an online platform so that it can be delivered virtually. We will also be integrated interpersonal aggression content to expand the logic and program theory of KIR to apply to situations in which violence may arise. The goal is to both delay initiation of AOD use/aggressive behaviors and change the youth's norms around the appropriateness of AOD use and interpersonal aggression. The intervention will delivered for the pilot study by members of the research team (PI and/or GRAs). The intervention materials will be translated into Spanish by a research team member who is a native speaker of Spanish and checked for accuracy by other members of team. Adaptations will be made in consultation with a community advisory board that consists of Venezuelan migrants to check for cultural fit, language appropriateness, and overall concordance with the target population. All members of the research team are either fluent or proficient in Spanish.

A three-armed RCT design will be used. In addition to a control group that will receive an abbreviated, one-session workshop, one group will receive a version of the intervention that has been adapted for Venezuelan youths and the other will receive a version of the intervention that has been adapted for Venezuelan youths and includes interpersonal violence content. The purpose of this design is to determine the effectiveness of the the culturally adaption of KiR for the original intended outcome (reduced AOD use) and the separate effect of integrating interpersonal violence content on reducing aggressive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Born in Venezuela
* Residing in U.S.
* Within age range

Exclusion Criteria:

* Substance use and/or engagement in interpersonal aggression will not be considered for purposes of inclusion/exclusion, unless the participant is intoxicated to the point of being unable to successfully complete a survey or participate in the intervention.
* Participants will be excluded if they are otherwise cognitively unable to successfully engage in the intervention

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Salas-Wright, PhD, Principal Investigator — Boston College
Locations (1):
- Raices Venezolanas, Doral, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- kiR + Aggression: The standard keepin' it REAL intervention was adapted for an online format, and there was content on interpersonal aggression. There was a 5-week and a 10-week version.
  kiR venezolano: A multi-week intervention focused on drug refusal skills and self-regulation.
Period: Overall Study
Arm/Group | Keepin' it REAL (kiR) | kiR + Aggression | Stress Management
Started | 12 | 14 | 8
Completed | 9 | 9 | 8
Not Completed | 3 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Keepin' it REAL (kiR) | kiR + Aggression | Stress Management | Total
Number analyzed (Participants) | 12 | 14 | 8 | 34
Age, Categorical [Count of Participants; unit: Participants] — Population: There were three groups involved in the trial.
  Participants
    <=18 years | 12 | 14 | 8 | 34
    Between 18 and 65 years | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We had three different arms in the trial.
  Participants
    Female | 6 | 5 | 6 | 17
    Male | 6 | 9 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Our trial had three arms.
  Participants
    Hispanic or Latino | 12 | 14 | 8 | 34
    Not Hispanic or Latino | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With No Alcohol Use
Description: We used one survey item from the self-report measure of substance use in prevention research scale, which asks youth how many alcoholic beverages they have consumed in the previous 30 days. Response options include none, only sips, all or part of one drink, 2 to 4 drinks, five to ten drinks, eleven to twenty drinks, and more than twenty drinks. No alcohol use ("none") during the study was considered a better outcome. There are no subscales or computed scores.
Time Frame: 3 months
Population: Participants who completed the baseline and 3-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Keepin' it REAL (kiR) | kiR + Aggression | Stress Management
Number analyzed (Participants) | 3 | 1 | 0
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With No Engagement in Interpersonal Aggression
Description: We used a composite scale of six items from the Revised Olweus Bully/Victim Questionnaire. The scale items measure the frequency of bullying activities, including making fun of, excluding, hitting, spreading rumors, threatening, and hurting others. Each item's responses include "almost never or never" (coded as 0), "weekly" (coded as 1), "several times per week" (coded as 2), and "daily" (coded as 3). Report of no bullying ("almost never or never") throughout the study was considered a better outcome.
Time Frame: 3 months
Population: Participants who completed baseline and three month follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Keepin' it REAL (kiR) | kiR + Aggression | Stress Management
Number analyzed (Participants) | 3 | 1 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Keepin' it REAL (kiR) | kiR + Aggression | Stress Management
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT05240313/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT05240313/SAP_001.pdf
  • Informed Consent Form (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT05240313/ICF_002.pdf